CLINICAL TRIAL: NCT02238782
Title: A Study to Assess the Absolute Bioavailability of a Single Oral Dose of Selumetinib With Respect to an Intravenous Microdose of [14C] Selumetinib in Healthy Male Volunteers
Brief Title: A Study to Assess the Absolute Bioavailability of Oral Selumetinib in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00080
Record Dates: First submitted 2014-08-08; First posted 2014-09-12 (Estimated); Results first posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteers Bioavailability Study
Keywords: bioavailability; pharmacokinetics; I phase; AZD6244; cancer
MeSH Terms: conditions — Neoplasms | interventions — AZD 6244

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- selumetinib 75mg single dose (Experimental): 3 capsules of 25 mg administered orally
  Interventions: Drug: selumetinib 75mg single dose; Other: [14C] selumetinib IV solution

INTERVENTIONS:
Drug: selumetinib 75mg single dose — 3 capsules of 25 mg given as a single dose
  Other Names: Selumetinib
Other: [14C] selumetinib IV solution — single, radiolabeled, IV (infused), microdose (80 μg) of [14C] selumetinib, infused using a syringe pump as a 15-minute infusion, administered 1h 15 min after receiving the oral dose

SUMMARY:
To assess the absolute bioavailability of oral selumetinib in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Healthy male volunteers aged 18 to 65
3. Male volunteers with sexual partners who are pregnant or who could become pregnant should use two highly effective methods of contraception (including one barrier method) for at least 14 days after completing the study and should avoid sperm donation for 14 days after study completion.
4. Body mass index between 18 and 30 kg/m2 and weighing between 50 and 100 kg.
5. Use no nicotine containing products for at least 3 months prior to screening with a negative cotinine screen at screening and Day 1 (Visit 2)
6. Calculated creatinine clearance greater than 50 mL/min using Cockcroft Gault formula.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study
2. Previous enrolment for treatment in the present study
3. Japanese or non Japanese Asian or Indian ethnicity.
4. Any one parent or grandparent is Japanese or non-Japanese Asian or Indian.
5. Treatment with another new chemical entity or participation in any other clinical study that included drug treatment within at least 3 months
6. Participation in another clinical study involving administration of [14C] radioactivity within 1 year.
7. Current or past history of central serious retinopathy or retinal vein thrombosis, intraocular pressure greater than 21 mmHg or uncontrolled glaucoma.
8. Any clinically significant disease or disorder which, may put the volunteer at risk because of participation in the study, influence the study result or influence the volunteer's ability to participate in the study.
9. Any clinically relevant abnormal findings in physical examination, haematology, clinical chemistry, urinalysis, vital signs or 12 lead ECG at Visit 1, which may put the volunteer at risk because of his participation in the study.
10. Use of drugs with enzyme inducing properties such as St John's Wort within 4 weeks prior to the administration of the investigational product
11. Use of any other prescribed medicine and over the counter drugs within 2 week or 5 times the half life, whichever is longer prior to the administration of the investigational product up to and including the follow up visit (Visit 4), with the exception of occasional use of paracetamol or ibuprofen and over the counter adrenergic nasal spray. No medications known to prolong the QT/corrected QT interval are allowed.
12. Excessive intake of caffeine containing drinks or food
13. Any intake of grapefruit and Seville oranges including products containing grapefruit or Seville oranges within 7 days of the admission on Day -1.
14. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to Selumetinib.
15. Plasma donation within 1 month of screening (Visit 1) or any blood donation or blood loss greater than 500 mL during the 3 months prior to screening (Visit 1).
16. History of or current alcohol or drug abuse.
17. A suspected or manifested infection according to the International Air Transport Association Categories A and B infectious substances.
18. Positive results on screening tests for HIV and/or hepatitis B and/or hepatitis C.
19. Baseline LVEF <55% measured by echocardiography.
20. Planned inpatient surgery, dental procedure or hospitalisation during the study.
21. Healthy male volunteers who in the opinion of the Principal Investigator, should not participate in the study.
22. Judgment by Principal Investigator that the volunteer should not participate in the study if they have ongoing or recent minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Research Site, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 21 subjects were enrolled, 12 of these subjects went on to receive treatment
Groups:
- Selumetinib: Patients received a single oral dose of selumetinib 75mg followed by IV carbon 14 selumetinib (80 micrograms) 1 hour 15 minutes after receiving the oral dose.
Period: Overall Study
Arm/Group | Selumetinib
Started | 12
Subjects Treated | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Selumetinib
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Absolute Bioavailability
Description: To calculate absolute bioavailability we used the formula: Area Under the Curve (oral dose)/Area Under the Curve (intravenous dose)*100
Time Frame: 0 to 72 hours post-dose
Measure: Geometric Mean (90% Confidence Interval); unit: % of bioavailability
Groups:
- Selumetinib: Selumetinib 75 mg oral followed by IV carbon 14 selumetinib (80 micrograms) administered 1 hour 15 minutes after the oral dose.
Arm/Group | Selumetinib
Number analyzed (Participants) | 12
% of bioavailability | 62.1 [60.1 to 64.1]

ADVERSE EVENTS:
Arm/Group | Selumetinib
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selumetinib (N=12)
Head Ache (Nervous system disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No